CLINICAL TRIAL: NCT02802280
Title: Personalized Medicine in HCV Chronic Infection. Endothelial Dysfunction and Subclinical Atheromatosis in Patients With HCV Infection. Characterization and Potential Reversibility With Direct Antiviral Agents.
Brief Title: Endothelial Dysfunction and Subclinical Atheromatosis in Chronic HCV Infection. Response to DAA Agents.
Acronym: C-Endys
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C-Endys PI15/02138; PI15/02138 (Other Grant/Funding Number: Spanish Ministry of Economy and Competitiveness)
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C; Cardiovascular Diseases
Keywords: endothelial dysfunction
MeSH Terms: conditions — Hepatitis C; Cardiovascular Diseases | interventions — Heart Disease Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular risk in HCV patients (Other): Intervention:
  The only intervention to be carried out along the study will consist of a complete evaluation of cardiovascular risk of HCV patients both at baseline (pre-treatment) and after HCV treatment, through performing different tests (see below)
  Chronic HCV patients who are going to be treated with new DAAs according to current guidelines will be studied at different times before and after the end of the treatment.
  The participation in the study will not influence neither the indication to treat nor the treatment used.
  Anti-HCV regimens will be used according to clinical practice as indicated into the current guidelines
  Interventions: Other: Cardiovascular risk in HCV patients

INTERVENTIONS:
Other: Cardiovascular risk in HCV patients — Cardiovascular risk assessement (through Flow-mediated vasodilatation "FMV", measurement of endothelial function biomarkers, carotid ultrasound, etc.)
  This is a prospective study. The only intervention planned will consist of performing different tests that define the individual cardiovascular risk. These tests will be carried out on a single group cohort at different times.
  Notwithstanding, the investigators will record the exposure to DAA to assess any change in CVR.
  Anti-HCV regimens will be used according to clinical practice as indicated into the current guidelines (1)
  (1)European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. PubMed PMID: 25911336.

SUMMARY:
Hypothesis: In addition to the liver deleterious effects, Chronic Hepatitis C (CHC) can cause changes in other organs highlighting the increased cardiovascular risk (CVR) through accelerated atherosclerosis, whose consequences may persist even after healing infection with new antiviral treatments. This can have major impact on the health system. Obtaining a Sustained Virological Response (SVR) with a free Interferon (IFN) antiviral treatment is probably able to reverse, at least partially, increased vascular risk induced by Hepatitis C virus (HCV) and perhaps ultimately reverse the subclinical atherosclerosis.

Aims: To study the presence of early-subclinical atherosclerotic disease (endothelial dysfunction and subclinical atherosclerosis) in patients with CHC and evaluate the influence of treatment in the short and medium term on the CVR derived. Studying these same issues but in patients with established atherosclerotic disease.

DETAILED DESCRIPTION:
Design:

Prospective interventional study.

Patients and methods:

Tracked on a population of 80 patients with CHC (estimated fibrosis F2-F3),

An evaluation of the CVR will be performed by determining biomarkers of endothelial activation and macrophage activation, measuring flow-mediated vasodilation and atherosclerotic damage.

All evaluations will take place prior (at baseline) and after antiviral treatment. Particularly, all determinations will be performed immediately before and 3, 12 and 24 months after the end of antiviral treatment.

In order to improve the diagnostic accuracy in terms of discriminating liver damage associated to Non Alcoholic Fatty Liver Disease (NAFLD) from HCV infection, the investigators will use the owl-liver® technique in all patients before and after treatment.

Sample size: Considering the primary endpoint the flow-mediated vasodilation (FMD), data have been reported on FMD of 7.6 ± 2.4% in healthy subjects and 5.1 ± 2.2% in subjects with risk factors (Dalli et al Rev Esp Cardiol 2002; 55: 928-35). Assuming these SD and a correlation coefficient of 0.3 between the two measurements, 80 patients will be needed to detect a change of 1% in vasodilation with an output of 90% and a significance level of 5%.

Variables and tasks:

Task 1. Assessment of endothelial function.

1. -Vasodilation mediated by ultrasound brachial flow through the rate of increase of brachial artery diameter (d2) as compared to baseline (d1) after a ischemia time (300 mmHg) for 4 minutes (FMD = (d2-d1) / d1 (x 100).
2. -Endothelial function biomarkers: ICAM-1, VCAM-1, E-selectin, P-selectin, MCP-1, angiopoietin-2, sTWEAK and ADMA.
3. - Macrophage activation biomarkers: Gal-3BP, sCD163 and sCD14.

Task 2. Assessment of atherosclerotic damage. Common carotid, internal carotid and carotid bulb (bilateral) will be explored by ultrasound. The images will be electronically stored in DICOM format.

The analyzed parameters will be:

1. cIMT (Carotid intima media thickness and carotid intima-media thickness) defined as the distance between the interface of the carotid lumen with arterial intima and the interface of medium with adventitia of the distal arterial wall. They will be measured on the back wall in a free-plaque area in the common carotid (cIMT CC) in the carotid bulb (cIMT -B), and internal carotid (cIMT -CI).
2. Presence of carotid plaques in these territories. Plaque will be defined following the Mannheim criteria.
3. Presence of atherosclerotic plaque: to distinguish between focal and diffuse thickening. In the focal plate area, maximum thickness and Gray Scale Median (GSM) will be quantified. In the diffuse thickening (IMT> 1.5 mm) only the GSM will be quantified.

Task 3. Assessment of vascular risk. Classic and emerging vascular risk assessment.

1. -Study of classic risk factors: through REGICOR and Framingham Score tables. Fatty Liver Index to exclude or confirm NASH (BMI, waist circumference, triglycerides and GGT). Metabolic syndrome will be detected by the NCEP-ATPIII.
2. - Study of emerging vascular risk factors, including proinflammatory factors. In this way, the investigators will analyze the plasma levels hcPCR, homocysteine, Lp(a), pentraxin 3, SAA, oxidized LDL, PON1, PCSK9 and elevated plasma levels of von Willebrand factor factor (VWF)
3. - Qualitative lipoprotein changes: the total concentration of lipoprotein (VLDL, LDL, HDL) will be determined as well as their composition (total cholesterol, triglycerides, phospholipids, protein, apolipoprotein B, lipoprotein ratio / total triglyceride mass VLDL, LDL and HDL, number of VLDL, LDL and HDL, cholesterol molecules per particle and triglyceride molecules per particle).
4. - Insulin resistance by HOMA.
5. -HbA1c
6. - Rx Thorax.

h)-ECG with QTc interval measurement.

ELIGIBILITY:
Inclusion Criteria:

* HCV infected patients (aged 18-75 yr)
* Naive or failure to previous treatments
* Liver fibrosis F2-F3 in Fibroscan/liver biopsy
* Accept the study and sign the CI

Exclusion Criteria:

* Known cardiovascular diseases
* Does not meet the above criteria
* VIH or other viral coinfection
* Hepatocarcinoma
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Flow mediated dilatation (FMD) | Basal and 3, 12 and 24 months after the end of treatment
  FMD: Vasodilation mediated by ultrasound brachial flow through the rate of increase of brachial artery diameter (d2) as compared to baseline (d1) after a ischemia time (300 mmHg) for 4 minutes (FMD = (d2-d1) / d1 (x 100).

SECONDARY OUTCOMES:
Changes in cIMT (Carotid intima-media thickness) | Basal and 3, 12 and 24 months after the end of treatment
  cIMT (Carotid intima-media thickness) will be assessed by carotid ultrasound. It is defined as the distance between the interface of the carotid lumen with arterial intima and the interface of medium with adventitia of the distal arterial wall. They will be measured on the back wall in a free-plaque area in the common carotid (cIMT CC) in the carotid bulb (cIMT -B), and internal carotid (cIMT -CI).
Changes in the presence of carotid plaques | Basal and 3, 12 and 24 months after the end of treatment
  Presence of carotid plaques in these territories (common carotid, carotid bulb and internal carotid). Plaque will be defined following the Mannheim criteria. It will be assessed by carotid ultrasound image.
Changes in ICAM-1 serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of ICAM-1 (Intercellular Adhesion Molecule 1) serum levels at different times (see time frame)
Changes in VCAM-1 serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of Vascular cell adhesion molecule 1 (VCAM-1) serum levels at different times (see time frame)
Changes in E-selectin serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of E-selectin serum levels at different times (see time frame)
Changes in P-selectin serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of P-selectin serum levels at different times (see time frame)
Changes in MCP-1 serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of monocyte chemoattractant protein 1 (MCP-1) serum levels at different times (see time frame)
Changes in galectin-3-binding protein serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of galectin-3-binding protein serum levels at different times (see time frame)
Changes in CD163 serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of CD163 (Cluster of Differentiation 163) serum levels at different times (see time frame)
Changes in hs-PCR serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of hs-PCR serum levels at different times (see time frame)
Changes in Lp(a) serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of Lipoprotein(a) (Lp(a)) serum levels at different times (see time frame)
Changes in VLDL serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of VLDL serum levels at different times (see time frame)
Changes in LDL serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of LDL serum levels at different times (see time frame)
Changes in HDL serum levels | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of HDL serum levels at different times (see time frame)
Changes in HOMA | Basal and 3, 12 and 24 months after the end of treatment
  Measurement of HOMA (homeostasis model assessment) index at different times (see time frame)
Presence of Sustained Viral Response | 3, 6 and 12 months after the end of treatment
  Data on efficacy of treatment
Adverse events | up to 24 weeks
  Data on safety of treatments

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crespo García, MDPhD, Principal Investigator — Head of Gastroenterology and Hepatology at Hospital Universitario Marqués de Valdecilla. Professor at the Universidad de Cantabria
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. No abstract available. PMID 25911336
- [Background] Petta S, Macaluso FS, Craxi A. Cardiovascular diseases and HCV infection: a simple association or more? Gut. 2014 Mar;63(3):369-75. doi: 10.1136/gutjnl-2013-306102. Epub 2013 Dec 2. No abstract available. PMID 24295849
- [Background] Negro F. Facts and fictions of HCV and comorbidities: steatosis, diabetes mellitus, and cardiovascular diseases. J Hepatol. 2014 Nov;61(1 Suppl):S69-78. doi: 10.1016/j.jhep.2014.08.003. Epub 2014 Nov 3. PMID 25443347
- [Background] Perticone M, Maio R, Tassone EJ, Tripepi G, Di Cello S, Miceli S, Caroleo B, Sciacqua A, Licata A, Sesti G, Perticone F. Insulin-resistance HCV infection-related affects vascular stiffness in normotensives. Atherosclerosis. 2015 Jan;238(1):108-12. doi: 10.1016/j.atherosclerosis.2014.11.025. Epub 2014 Nov 29. PMID 25461736